CLINICAL TRIAL: NCT06484907
Title: Predictive Power of the ACTA-PORT Score for Cardiac Surgery-Associated Acute Kidney Injury: A Prospective Observational Study
Brief Title: Predicting CSA-AKI With ACTA-PORT Score
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Cansuhan AKAR YİĞİT, Assistant Doctor, Ankara City Hospital Bilkent
Other Study IDs: ABCH-AR-CAY-01
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Disease; Blood Transfusion; Acute Kidney Injury
Keywords: Cardiopulmonary Bypass; Cardiac Surgery; Transfusion; Acute Kidney Injury; ACTA PORT
MeSH Terms: conditions — Heart Diseases; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In the scope of this study, it will be determined whether the ACTA-PORT (Association of Cardiothoracic Anesthetists perioperative risk of blood transfusion) scoring system can predict the incidence of events in other organ systems, and the feasibility of conducting multiple assessments using a single simple score will be investigated.

DETAILED DESCRIPTION:
ACTA-PORT (Association of Cardiothoracic Anesthetists perioperative risk of blood transfusion) score is a simple, reliable, and validated tool used to predict the risk of transfusion in patients undergoing heart surgery. In calculating ACTA-PORT score, age, gender, hemoglobin, body surface area, EuroSCORE, creatinine, and type of operation are used.

In this study, it will be determined whether the ACTA-PORT (Association of Cardiothoracic Anesthetists perioperative risk of blood transfusion) scoring system can predict the incidence of events in other organ systems, and the feasibility of conducting multiple assessments using a single simple score will be investigated.

The files of patients undergoing open heart surgery in the cardiovascular surgical operating rooms of Ankara Bilkent City Hospital, along with anesthesia records, transfusion records, and test results identified through the Hospital Information Management System, will be prospectively evaluated. Data will be collected after patients are admitted to the intraoperative and postoperative intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients having open heart surgery
* Patients undergoing surgery by using cardiopulmonary bypass pump

Exclusion Criteria:

* Patients under 18 years old
* Patients diagnosed with kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having open heart surgery by using cardiopulmonary bypass pump in Ankara Bilkent City Hospital between 01 July 2024 - 01 November 2024.
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
KDIGO AKI Staging | Preoperative (last week before operation) and daily after the operation for 7 days
  KDIGO is in the process of developing the Clinical Practice Guideline for Acute Kidney Injury (AKI) and Acute Kidney Disease (AKD). ///// Stage 1: Serum creatinine 1.5-1.9 times baseline or ≥0.3 mg/dl (≥26.5 mmol/l) increase or Urine output <0.5 ml/kg/h for 6-12 hours ////// Stage 2: Serum creatinine 2.0-2.9 times baseline or <0.5 ml/kg/h for ≥12 hours /////// Stage 3: Serum creatinine 3.0 times baseline or Increase in serum creatinine to ≥4.0 mg/dl (≥353.6 mmol/l) or Initiation of renal replacement therapy or in patients <18 years, decrease in eGFR to <35 ml/min per 1.73 m² or Urine output <0.3 ml/kg/h for ≥24 hours or anuria for ≥12 hours

SECONDARY OUTCOMES:
Mechanical Ventilation Duration | the duration after surgery up to a month
  The duration the patient remains intubated from surgery to extubation
Intensive Care Duration | the duration after surgery up to a month
  The duration the patient remains in intensive care unit after surgery
Hospital Stay Duration | the duration after surgery up to a month
  The duration the patient stays in the hospital after surgery until discharge
Mortality | the duration after surgery up to a month
  If the patient dies within 1 month or not
Complications | the duration after surgery up to a month
  Cardiac, Pulmonary, Neurological, Infectious, Thrombotic complications and Presence of MODS (Multiple Organ Dysfunction Syndrome) / SIRS (Systemic Inflammatory Response Syndrome)
Reoperation Necessity | the duration after surgery up to a month
  The need for reoperation due to bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Asli DEMIR, Ph.D, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No